CLINICAL TRIAL: NCT03349008
Title: The Efficacy and Safety Study of Magnesium Isoglycyrrhizinate Injection Followed by Diammonium Glycyrrhizinate Enteric-coated Capsules and Combined With Entecavir on the Treatment of Chronic Hepatitis B
Brief Title: Magnesium Isoglycyrrhizinate Followed by Diammonium Glycyrrhizinate and Combined With Entecavir in Chronic Hepatitis B
Acronym: MAGIC-101
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cttq (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cttq-MAGIC-101
Record Dates: First submitted 2017-05-04; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Chronic Hepatitis b; Liver Inflammation
Keywords: necro-inflammatory; glycyrrhizin; entecavir; hepatic biological parameters; liver fibrosis
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis; Liver Cirrhosis | interventions — entecavir; 18alpha,20beta-hydroxy-11-oxo-norolean-12-en-3beta-yl-2-O-beta-D-glucopyranurosyl-alpha-D-glucopyranosiduronate magnesium tetrahydrate; Glycyrrhizic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Entecavir treatment with placebo, Magnesium Isoglycyrrhizinate placebo followed by Diammonium Glycyrrhizinate placebo
  Interventions: Drug: Entecavir; Drug: Magnesium Isoglycyrrhizinate Placebo; Drug: Diammonium Glycyrrhizinate Placebo
- Experimental group (Experimental): Entecavir combined with glycyrrhizin, Magnesium Isoglycyrrhizinate Injection followed by Diammonium Glycyrrhizinate
  Interventions: Drug: Entecavir; Drug: Magnesium Isoglycyrrhizinate; Drug: Diammonium Glycyrrhizinate

INTERVENTIONS:
Drug: Entecavir — Glycyrrhizin for the treatment of patients with chronic hepatitis B combined with entecavir-based
  Other Names: Entecavir Pill
Drug: Magnesium Isoglycyrrhizinate — Magnesium Isoglycyrrhizinate Injection treat for two weeks with entecavir-based
  Other Names: Magnesium Isoglycyrrhizinate Injection
  Arms: Experimental group
Drug: Diammonium Glycyrrhizinate — Diammonium Glycyrrhizinate for oral after Magnesium Isoglycyrrhizinate Injection treatment with entecavir-based
  Other Names: Diammonium Glycyrrhizinate Enteric-coated Capsules
  Arms: Experimental group
Drug: Magnesium Isoglycyrrhizinate Placebo — Magnesium Isoglycyrrhizinate Injection Placebo
  Other Names: Magnesium Isoglycyrrhizinate Injection Placebo
  Arms: Control group
Drug: Diammonium Glycyrrhizinate Placebo — Diammonium Glycyrrhizinate Enteric-coated Capsules Placebo
  Other Names: Diammonium Glycyrrhizinate Enteric-coated Capsules Placebo
  Arms: Control group

SUMMARY:
This study evaluates the addition of glycyrrhizin to entecavir in the treatment of patients with chronic hepatitis B in China. Half of participants will receive magnesium isoglycyrrhizinate followed by oral diammonium glycyrrhizinate and entecavir in combination, while the other half will receive a placebo and entecavir.

DETAILED DESCRIPTION:
Chronic hepatitis B(HBV) has a high prevalence (>8%) in China. Entecavir, aguanosine analog, is a potent and selective inhibitor of HBV DNA polymerase.

Glycyrrhizin has been used for more than 30 years in the treatment of liver diseases in Asian countries, who can relieve necro-inflammatory and liver fibrosis or cirrhosis Recent study has shown that inflammation plays the important role in chronic HBV and fibrosis or cirrhosis disease progression, but antiviral therapy only may not reduce inflammation ideally. The addition of glycyrrhizin to entecavir in the treatment may slow disease progression in patients with chronic HBV and advanced fibrosis or cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis B surface antigen [HBsAg]-positive,
* Either hepatitis B e antigen (HBeAg)-positive or HBeAgnegative/hepatitis B e antibody (HBeAb)-positive disease were eligible,
* Serum alanine aminotransferase (ALT) levels 3-10×the upper limit of normal (ULN),serum total bilirubin(TBIL)levels<2×ULN

Exclusion Criteria:

* Co-infection with hepatitis C virus, hepatitis D virus, or human immunodeficiency virus;
* Other forms of liver disease;
* More than 24 weeks of therapy with a nucleoside or nucleotide analog with activity against HBV, and therapy with any anti-HBV drug within 24 weeks prior to randomization;
* More than 12 weeks of therapy with liver protectants, and therapy with glycyrrhizin;
* Has decompensated liver function or has a hint of hepatocellular carcinoma (HCC);
* During the study patients were not allowed to use other medicines.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2017-11-25 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of ALT(Alanine aminotransferase) | baseline and 24 weeks
  The ALT levels of plasma are measured at baseline and at 24 weeks. The normal value was 0-40 U/L.

SECONDARY OUTCOMES:
Change of Liver inflammatory | baseline and 24 weeks
  Liver inflammatory of the liver biopsies is performed at baseline and 24 weeks evaluated by Knodell HAI score.
Change of Liver Fibrosis | baseline and 96 weeks
  Liver Fibrosis is performed at baseline and 96 weeks evaluated by Fibroscan examination.

IPD SHARING:
Plan to Share IPD: Undecided